CLINICAL TRIAL: NCT02890433
Title: Are Standard Precautions as Efficient as Contact Additional Precautions Against the Transmission of Multi-drug Resistant Bacteria in Intensive Care Unit ?
Brief Title: Standard Precautions Versus Contact Additional Precautions Against Multi-drug Resistant Bacteria in Intensive Care Unit (PSBMR)
Acronym: PSBMR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-06Obs-CHRMT
Record Dates: First submitted 2016-08-26; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Multi-drug Resistant Bacteria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The national recommendations promote the applying of the Contact Additional Precautions (CAP) with the Standard Precautions (SP) to limit the transmission of multi-drug resistant (MDR) bacteria. However, that could entail more costs and a reduction of quality of the patient care.

DETAILED DESCRIPTION:
The national recommendations promote the applying of the Contact Additional Precautions (CAP) with the Standard Precautions (SP) to limit the transmission of multi-drug resistant (MDR) bacteria. However, that could entail more costs and a reduction of quality of the patient care.

This study seeks showing it in way of a non-interventional research in a resuscitation unit. Two periods are compared for noticing the rates of MDR bacteria contaminations.

ELIGIBILITY:
Inclusion Criteria:

* hospitalization in resuscitation unit

Exclusion Criteria:

* opposition for gathering data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients hospitalized in the resuscitation unit of the study
Sampling Method: Non-Probability Sample
Enrollment: 3124 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Rate of Meticillin Resistant Staphylococcus Aureus (MRSA) and Enterobacteriaceae producing Extended Spectrum Beta-Lactamase (EESBL) per 1000 hospitalization days | 1000 days

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne SELLIES, MD, Principal Investigator — CHR Metz-Thionville
Locations (1):
- CHR Metz-Thionville, Metz, France